CLINICAL TRIAL: NCT00795093
Title: Partial Response to PPI Treatment: The Cost to Society and the Burden to the Patient
Brief Title: Partial Response to Proton Pump Inhibitors (PPI) Treatment: The Cost to Society and the Burden to the Patient - a Study in the US
Acronym: REMAIN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: i3 Innovus (Industry)
Responsible Party: Debra Silberg, MD PhD, Medical Science Director, Clinical Research, AstraZeneca R&D
Other Study IDs: D9120N00005
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2010-05

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GERD; PPI; partial responders
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: 552 GERD patients, partial responders to PPI treatment

SUMMARY:
The purpose of this study is to describe common treatment pathways, to collect health care utilization data and to assess symptom load as well as impact of symptoms on daily life in GERD patients who are partial-responders to PPI treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 month history of GERD symptoms
* Treated with unchanged optimized PPI treatment for any GERD indication during a consecutive 4 week period
* Remaining GERD symptoms despite optimized PPI treatment
* Able to read and write in US English, and able to comply with study requirements

Exclusion Criteria:

* Patients that have not experienced any GERD symptom improvement at all during PPI treatment
* Involvement in the planning or conduct of the study
* Involvement in any other observational study or in any clinical study at the time of this study or during the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Gastroesophageal Reflux Disease (GERD) classified as partial responders to proton pump inhibitors (PPIs).
Sampling Method: Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Quality of life, productivity loss, frequency and severity of GERD symptoms, health care resource use | Collected at enrollment visit and at 3 and 6 month follow-up. (Health care resource use is at enrollment visit collected retrospectively 6 months)
Utility values | Collected at enrollment visit and at 6 month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Meg Good, Principal Investigator — i3 Innovus; Marie Sundin, Study Director — AstraZeneca
Locations (53):
- United States (53):
  - Research Site, Leeds, Alabama
  - Research Site, Pheonix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Concord, California
  - Research Site, Lancaster, California
  - Research Site, Los Banos, California
  - Research Site, Solana Beach, California
  - Research Site, Newark, Delaware
  - Research Site, Altamonte Springs, Florida
  - Research Site, Cocoa, Florida
  - Research Site, DeFuniak Springs, Florida
  - Research Site, Largo, Florida
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Peonia, Florida
  - Research Site, Tampa, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Royston, Georgia
  - Research Site, Snellville, Georgia
  - Research Site, Belleville, Illinois
  - Research Site, Mishawaka, Indiana
  - Research Site, Metaire, Louisiana
  - Research Site, Prince Frederick, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Florissant, Missouri
  - Research Site, Jefferson City, Missouri
  - Research Site, Atco, New Jersey
  - Research Site, Fair Lawn, New Jersey
  - Research Site, Cary, North Carolina
  - Research Site, Elkin, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Stanley, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Beachwood, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Vandalia, Ohio
  - Research Site, Aliquippa, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Athens, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Irving, Texas
  - Research Site, San Antonio, Texas
  - Research Site, San Marcos, Texas
  - Research Site, Southlake, Texas
  - Research Site, West Jordan, Utah